CLINICAL TRIAL: NCT01706120
Title: A MULTICENTER STUDY IN PATIENTS WITH STAGE III-IV EPITHELIAL OVARIAN CANCER TREATED WITH CARBOPLATIN/PACLITAXEL WITH BEVACIZUMAB: CLINICAL AND BIOLOGICAL PROGNOSTIC FACTORS
Brief Title: Study of Clinical and Biological Prognostic Factors in Patients With Ovarian Cancer Receiving Carboplatin +Paclitaxel With Bevacizumab
Acronym: MITO16/MANGO-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITO-16 - MANGO-OV2; 2012-003043-29 (EudraCT Number)
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: prognostic factors; biologic factors; clinical factors; routine clinical practice
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- First-line chemotherapy with bevacizumab (Other): * Bevacizumab 15 mg/kg i.v. on Day 1 every 3 weeks for up to 22 cycles
  * Paclitaxel 175 mg/m2 on Day 1 every 3 weeks for up to 6 cycles
  * Carboplatin (AUC 5) on Day 1 every 3 weeks for up to 6 cycles
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Bevacizumab — • Bevacizumab 15 mg/kg i.v. on Day 1 every 3 weeks up to 22 cycles
  Other Names: Avastin
Drug: Paclitaxel — • Bevacizumab 15 mg/kg i.v. on Day 1 every 3 weeks up to 6 cycles
Drug: Carboplatin — • Carboplatin (AUC 5) on Day 1 every 3 weeks for up to 6 cycles

SUMMARY:
The addition of bevacizumab to first-line chemotherapy has been shown to improve progression free survival for patients with ovarian cancer. The purpose of this study is to explore the potential role of clinical and biologic factors in identifying those patients who benefit most from this combined therapy in terms of progression free and overall survival.

DETAILED DESCRIPTION:
MITO-16 - MANGO-OV2 is a single-arm, open-label, non-comparative, multicenter, phase IV study. Patients will receive a combination of bevacizumab, paclitaxel and carboplatin as first line treatment (in-label dose and scheduling). This is an exploratory study attempting to identify potential prognostic clinical factors(such as hypertension) and prognostic biologic factors. Overall, 2 types of biomarkers are considered. Dynamic biomarkers are those expressing the changing nature of the disease in relation to the treatment or simply the tumour progression, these are typically not inherited. Genetic biomarkers are typically inherited and are expression of some characteristics potentially able to interfere with the treatment effect (i.e. Pharmacogenomics).

The safety of this regimen in routine clinical practice will also be described.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥18 years of age.
* Patients with histologically confirmed epithelial ovarian carcinoma, fallopian tube carcinoma or primary peritoneal carcinoma, including mixed Mullerian Tumours Or Recurrent early stage epithelial ovarian or fallopian tube carcinoma treated with surgery alone.
* FIGO stage IIIB & C or IV
* ECOG Performance Status of 0-2.
* Life expectancy of at least 12 weeks.
* Signed informed consent obtained prior to initiation of any study-specific procedures and treatment as confirmation of the patient's awareness and willingness to comply with the study requirements.
* Availability of tumour samples for molecular analyses

Exclusion Criteria:

Cancer related

* Ovarian tumours with low malignant potential (i.e. borderline tumours)
* Previous systemic anti-cancer therapy for advanced ovarian cancer.
* History or evidence of brain metastases or spinal cord compression.
* History or evidence of synchronous primary endometrial carcinoma, unless all of the following criteria related to the endometrial carcinoma are met:

  * stage ≤Ia
  * no more than superficial myometrial invasion
  * no lymphovascular invasion
  * not poorly differentiated (grade 3 or papillary serous or clear cell carcinoma).
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.

Other-treatment related

* Any prior radiotherapy to the pelvis or abdomen.
* Surgery (including open biopsy) within 4 weeks prior to the first bevacizumab dose or planned (In this case the patient can be enrolled but the administration of bevacizumab should be omitted at first cycle).
* Current or recent (within 10 days prior to the first study drug dose) use of full-dose oral or parenteral anticoagulant or thrombolytic agent for therapeutic purposes (except for central venous access patency, in which case international normalized ratio [INR] must be maintained below 1.5). Post operative prophylaxis with low molecular weight heparin sc is allowed.
* Current or recent (within 30 days of first study dosing) treatment with another investigational drug.

Laboratory related

* Inadequate bone marrow function: ANC: <1.5 x 109/l, or platelet count <100 x 109/l or Haemoglobin <9 g/dl. Patients may be transfused to maintain haemoglobin values ≥9 g/dl.
* Inadequate coagulation parameters:

  * activated partial thromboplastin time (APTT) >1.5 xULN or
  * INR >1.5
* Inadequate liver function, defined as:

  * serum (total) bilirubin >1.5 x the upper limit of normal (ULN) for the institution
  * AST/SGOT or ALT/SGPT >2.5 x ULN.
* Inadequate renal function, defined as serum creatinine >2.0 mg/dl or >177 micromol/l
* Proteinuria >1g in a 24-hour urine collection (to be performed only among patients who showed a ≥3+ at urine dipstick).

Patient related

* Pregnant or lactating patients.
* History or evidence of thrombotic or hemorrhagic disorders; including cerebrovascular accident (CVA) / stroke or transient ischemic attack (TIA) or sub-arachnoid haemorrhage within ≤6 months prior to the first study treatment).
* Uncontrolled hypertension (sustained systolic >150 mm Hg and/or diastolic >100 mm Hg despite antihypertensive therapy) or clinically significant (i.e. active) cardiovascular disease, including:

  * myocardial infarction or unstable angina within ≤6 months prior to the first study treatment
  * New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF)
  * serious cardiac arrhythmia requiring medication (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia)
  * peripheral vascular disease ≥grade 3 (i.e. symptomatic and interfering with activities of daily living requiring repair or revision).
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to the first study treatment.
* Non-healing wound, ulcer or bone fracture. Patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require three weekly wound examinations.
* Evidence of any other medical conditions (such as psychiatric illness, peptic ulcer, etc.), physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-10; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
expression of soluble and tissutal biomarkers | measured at baseline, at completion of chemotherapy, at disease progression or bevacizumab completion up to 15 monthsfor each patient

SECONDARY OUTCOMES:
progression free survival | one year
overall survival | three years
worst grade toxicity per patient | evaluated every 3 weeks up to 15 month
  according to Common Toxicity Criteria for Adverse Events v. 4.03
number of patients taking oral antidiabetic therapy | at baseline
number of patients taking antithrombotic therapy | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Nicoletta Colombo, M.D., Principal Investigator — European Institute of Oncology; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Gennaro Daniele, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Roldano Fossati, M.D., Principal Investigator — Mario Negri Institute; Ciro Gallo, M.D., Principal Investigator — University of Campania Luigi Vanvitelli; Irene Floriani, Ph.D., Principal Investigator — Mario Negri Institute
Locations (47):
- Italy (47):
  - A.S.O. SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Centro di Riferimento Oncologico, Aviano
  - Ospedale Fatebenefratelli, Benevento
  - Spedali Civili - Università di Brescia, Brescia
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Fondazione del Piemonte per l'Oncologia, Candiolo
  - Ospedale Ramazzini di Carpi /Ospedale di Mirandola, Carpi
  - Azienda Ospedaliera Garibaldi Nesimadi Catania, Catania
  - Ospedale Cannizzaro, Catania
  - Ospedale Mater Domini, Catanzaro
  - Ospedale Civile di Faenza, Faenza
  - Ospedale Santa Croce, Fano
  - A.O.U. Arcispedale Sant'Anna di Ferrara, Ferrara
  - Ospedale Fabrizio Spaziani di Frosinone / Osp. SS Trinità di Sora, Frosinone
  - E.O. Ospedali Galliera, Genova
  - IRCCS San Martino IST, Genova
  - Ospedale di Guastalla, Guastalla
  - Ospedale A. Manzoni, Lecco
  - Ospedale Mater Salutis, Legnago
  - Presidio Ospedaliero Manerbio, Manerbio
  - A.O. C. Poma, Mantova
  - Istituto Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori, Milan
  - Ospedale San Raffaele, Milan
  - U.L.S.S. 13, Mirano
  - A.O.U. Policlinico Modena, Modena
  - Ospedale S. Gerardo, Monza
  - AOU Policlinico Federico II, Napoli
  - Istituto Nazionale dei Tumori, Napoli
  - Istituto Sacro Cuore Don Calabria, Negrar
  - Istituto Oncologico Veneto, Padua
  - Fondazione IRCCS S. Matteo, Pavia
  - Ospedale Silvestrini, Perugia
  - Ospedale Santa Chiara, Pisa
  - A.O. Santa Maria degli Angeli, Pordenone
  - Ospedale S. Maria delle Croci, Ravenna
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale degli Infermi / Ospedale Civile, Rimini
  - Istituto Regina Elena, Roma
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma
  - Policlinico Universitario Gemelli Università Cattolica del Sacro Cuore, Roma
  - A.O. Ordine Mauriziano, Torino
  - A.O.U. OIRM-S. Anna, Torino
  - ASS N 1 Triestina, Trieste
  - A.O. di Udine S. Maria delle Misericordia, Udine
  - Ospedale del Ponte, Varese

REFERENCES:
- [Derived] Di Liello R, Arenare L, Raspagliesi F, Scambia G, Pisano C, Colombo N, Frezzini S, Tognon G, Artioli G, Gadducci A, Lauria R, Ferrero A, Cinieri S, De Censi A, Breda E, Scollo P, De Giorgi U, Lissoni AA, Katsaros D, Lorusso D, Salutari V, Cecere SC, Lapresa M, Nardin M, Bogani G, Distefano M, Greggi S, Gargiulo P, Schettino C, Gallo C, Daniele G, Califano D, Perrone F, Pignata S, Piccirillo MC. Thromboembolic events and antithrombotic prophylaxis in advanced ovarian cancer patients treated with bevacizumab: secondary analysis of the phase IV MITO-16A/MaNGO-OV2A trial. Int J Gynecol Cancer. 2021 Oct;31(10):1348-1355. doi: 10.1136/ijgc-2021-002786. Epub 2021 Aug 30. PMID 34462317
- [Derived] Daniele G, Raspagliesi F, Scambia G, Pisano C, Colombo N, Frezzini S, Tognon G, Artioli G, Gadducci A, Lauria R, Ferrero A, Cinieri S, De Censi A, Breda E, Scollo P, De Giorgi U, Lissoni AA, Katsaros D, Lorusso D, Salutari V, Cecere SC, Zaccarelli E, Nardin M, Bogani G, Distefano M, Greggi S, Piccirillo MC, Fossati R, Giannone G, Arenare L, Gallo C, Perrone F, Pignata S. Bevacizumab, carboplatin, and paclitaxel in the first line treatment of advanced ovarian cancer patients: the phase IV MITO-16A/MaNGO-OV2A study. Int J Gynecol Cancer. 2021 Jun;31(6):875-882. doi: 10.1136/ijgc-2021-002434. Epub 2021 Apr 30. PMID 33931498